CLINICAL TRIAL: NCT05911984
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetic Properties and Preliminary Efficacy of 9MW3811 in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetic Properties and Preliminary Efficacy of 9MW3811 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW3811-2023-CP102
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9MW3811 Injection (Experimental)
  Interventions: Drug: 9MW3811 Injection

INTERVENTIONS:
Drug: 9MW3811 Injection — Intravenous injection

SUMMARY:
This is a single ascending dose study of 9MW3811, the primary objective of which is to evaluate the safety, tolerability and preliminary efficacy of 9MW3811 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 18 and 75 years of age, inclusive.
2. Histologically or cytologically confirmed advanced malignant solid tumors, for which standard therapy does not exist or has proven ineffective or intolerable.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 3 months.
5. Participants must have measurable disease according to RECIST (version 1.1).
6. Adequate organ functions.
7. Sexually active fertile participants, and their partners, must agree to use methods of contraception during the study and at least 6 months after termination of study therapy.

Exclusion Criteria:

1. Participants with cancerous meningitis and/or central nervous system metastases with clinical symptoms.
2. History of other active malignant tumor within 3 years prior to screening.
3. Suffering from poorly controlled body cavity effusion.
4. Suffering from active autoimmune disease.
5. History of chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, or other respiratory diseases that require hospitalization within 4 weeks prior to the first dose of study drug.
6. History of clinically significant cardiac or cerebrovascular diseases within 6 months prior to the first dose of study drug.
7. History of other severe or uncontrolled systemic disease, i.e. poorly controlled diabetes.
8. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
9. Major surgery within 28 days prior to the first dose of study drug.
10. Participants with one or more clinically significant positive test results of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, treponema pallidum antibody or human immunodeficiency virus (HIV) antibody.
11. Participants who have received treatment with biotherapy, endocrine therapy, immunotherapy, or other anti-tumor therapy within 2 weeks prior to the first dose of study drug; Radical radiotherapy received within 3 weeks or palliative radiotherapy received within 2 weeks prior to the first dose of study drug; Received treatment with chemotherapy within 3 weeks prior to the first dose of study drug (6 weeks for nitrosourea or mitomycin); Received treatment with oral fluorouracil or small molecule targeted drugs within 2 weeks or 5 half-lives prior to the first dose of study drug (whichever is shorter); Received treatment with anti-tumor traditional Chinese medicine within 1 week prior to the first dose of study drug; Participated in other clinical trials within 4 weeks prior to the first dose of study drug.
12. Participants who have received systemic treatment with immunosuppressants within 2 weeks prior to the first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) as assessed by CTCAE v5.0 | up to 24 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Incidence of dose-limiting toxicity (DLT) as assessed by CTCAE v5.0 | Cycle 1 Day 1 to Cycle 1 Day 21
  A DLT is defined as any of the adverse drug reactions listed in the protocol that will be assessed during Cycle 1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 evaluated by investigators | up to 24 weeks
  To determine the preliminary efficacy of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Disease Control Rate (DCR), According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 evaluated by investigators | up to 24 weeks
  To determine the preliminary efficacy of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Duration of Response (DoR), According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 evaluated by investigators | up to 24 weeks
  To determine the preliminary efficacy of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Progression Free Survival (PFS), According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 evaluated by investigators | up to 24 weeks
  To determine the preliminary efficacy of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Maximum Plasma Concentration (Cmax) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Time to reach Cmax (Tmax) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Terminal elimination half-life (t1/2) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
AUC from time 0 extrapolated to infinity (AUC0-inf) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Terminal elimination rate constant (λz) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Apparent clearance (CL) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Volume of distribution (Vz) | up to 24 weeks
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in patients with advanced solid tumors.
Incidence of antidrug antibodies (ADA) at specified timepoints relative to baseline | up to 24 weeks
  To determine the immunogenicity of 9MW3811.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No